CLINICAL TRIAL: NCT00027690
Title: A Phase II Trial of ZD 1839 (IRESSA) (NSC #715055) in the Treatment of Persistent or Recurrent Endometrial Carcinoma
Brief Title: Gefitinib in Treating Patients With Persistent or Recurrent Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Gynecologic Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02429; NCI-2012-02429 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000069057; GOG-0229C (Other: Gynecologic Oncology Group); GOG-0229C (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2001-12-07; First posted 2003-01-27 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Recurrent Uterine Corpus Carcinoma
MeSH Terms: interventions — Gefitinib

ARMS (1):
- Treatment (gefitinib) (Experimental): Patients receive oral gefitinib once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Gefitinib; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Gefitinib — Given orally
  Other Names: ZD 1839
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
Phase II trial to study the effectiveness of gefitinib in treating patients who have persistent or recurrent endometrial cancer. Biological therapies such as gefitinib may interfere with the growth of tumor cells and slow the growth of endometrial cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the 6-month progression-free survival of patients with persistent or recurrent endometrial carcinoma after receiving gefitinib.

II. Determine the nature and degree of toxicity of this drug in these patients. III. Determine the progression-free and overall survival of patients treated with this drug.

IV. Determine the effects of this drug on the levels of epidermal growth factor receptors (EGFR), c-ErbB2 (HER-2/neu) receptors, estrogen receptors (ER), and progesterone receptors (PR) (both PR and PRB) in tumor specimens of these patients.

V. Determine if an association exists between the levels of EGFR, ER, PR, PRB, and HER-2/neu serum concentrations of gefitinib, gefitinib activity, and soluble EGFR and clinical outcome in patients treated with this drug.

VI. Determine the frequency of clinical response (partial and complete response) in patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive oral gefitinib once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 22-60 patients will be accrued for this study within 2.5-6 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary endometrial carcinoma

  * Recurrent or persistent disease
* Received 1 prior chemotherapy regimen for endometrial carcinoma

  * Initial treatment may include high-dose, consolidation, or extended therapy administered after surgical or nonsurgical assessment
* At least 1 unidimensionally measurable lesion

  * At least 20 mm by conventional techniques (including palpation, plain x-ray, CT scan, and MRI)
  * At least 10 mm by spiral CT scan
  * Must have at least 1 target lesion for response assessment
  * Tumors within a previously irradiated field are designated as non-target lesions

    * Disease in a previously irradiated field as the only site of measurable disease is allowed only if there has been clear progression of the lesion since the completion of radiotherapy
* Must have a tumor that is accessible for guided core needle or fine needle biopsy
* Ineligible for a higher priority GOG protocol, defined as any active phase III protocol for the same patient population, if one exists
* Performance status - GOG 0-2 (for patients who received 1 prior regimen)
* Performance status - GOG 0-1 (for patients who received 2 prior regimens)
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN
* Creatinine no greater than 1.5 times ULN
* No unstable cardiac disease or myocardial infarction within the past 6 months
* History of coronary artery disease, congestive heart failure, or dysrhythmia allowed if on a stable regimen for at least 3 months
* No active infection requiring antibiotics
* No active corneal disease (e.g., keratoconjunctivitis)
* No grade 2 or greater sensory and motor neuropathy
* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer
* No signs or symptoms of bowel dysfunction that would preclude successful ingestion of oral study medication
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* At least 3 weeks since prior immunologic agents directed at malignant tumor
* No concurrent anticancer immunotherapy
* See Disease Characteristics
* At least 3 weeks since prior chemotherapy directed at the malignant tumor and recovered
* No prior non-cytotoxic chemotherapy for recurrent or persistent disease
* No concurrent anticancer chemotherapy
* At least 1 week since prior hormonal therapy directed at malignant tumor
* No concurrent anticancer hormonal therapy
* See Disease Characteristics
* At least 3 weeks since prior radiotherapy directed at malignant tumor and recovered
* No concurrent anticancer radiotherapy
* At least 4 weeks since prior surgery except minor procedures using local anesthesia (e.g., placement of a central venous port) and recovered
* At least 3 weeks since any other prior therapy directed at malignant tumor
* One additional prior cytotoxic regimen for recurrent or persistent disease allowed
* No prior gefitinib or other epidermal growth factor receptor inhibitor
* No prior cancer treatment that would contraindicate study therapy
* No concurrent CYP 3A4 inducers (including phenytoin, carbamazepine, barbiturates, nafcillin, rifampin, or Hypericum perforatum [St. John's Wort])
* No other concurrent investigational or antineoplastic agents
* No concurrent chlorpromazine

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2002-06; Primary Completion 2004-09 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients alive and progression-free | 6 months
Frequency and severity of adverse effects as assessed by National Cancer Institute Common Toxicity Criteria (CTC) v2.0 | Up to 5 years

SECONDARY OUTCOMES:
Duration of progression-free survival | Up to 5 years
Duration of overall survival | Up to 5 years
Frequency of clinical response utilizing the Gynecologic Oncology Group (GOG) Response Evaluation Criteria in Solid Tumors (RECIST) criteria | Up to 5 years
Numerical descriptions of serum concentrations of gefitinib, gefitinib activity, and soluble epidermal growth factor receptor (EGFR) | Baseline to end of course 5
Initial performance status and histological grade | Baseline to end of course 5

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Leslie, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States